CLINICAL TRIAL: NCT01878591
Title: Can Ultrasound Predict Labor Outcome in Operative Vaginal Deliveries?
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: St.Olavs Hospital, Trondheim University Hospital, Norway (Unknown); Lund University Hospital (Other); University of Bologna (Other); Copenhagen University Hospital, Hvidovre (Other); Queen Charlotte's and Chelsea Hospital (Other); University of Parma (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1865; 2012/186 (Other: REK-VEST)
Record Dates: First submitted 2013-06-09; First posted 2013-06-17 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Prolonged Labour
Keywords: labour; dystocia; operative delivery; vacuum; ultrasound
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women in active second stage of labour: Ultrasound examinations

SUMMARY:
To assess whether ultrasound methods can predict outcome of operative vaginal deliveries in nulliparous women at term with singleton pregnancies and prolonged second stage of labor.

To compare different ultrasound assessments Compare digital assessments and ultrasound findings. Investigate if movement of the fetal head during active pushing is a predictive factor

Null hypotheses:

* Ultrasound measurements cannot predict outcomes of operative vaginal delivery.
* Ultrasound is not better than digital examination in predicting delivery outcome.
* Movement of fetal head with active pushing is not a predictive factor.

DETAILED DESCRIPTION:
The physician responsible for the labor will perform digital examinations (fetal station and position and cervical dilatation). Fetal station will be related to the ischial spine from -5 to +4 as described by WHO and illustrated in Figure 111. Another obstetrician or midwife blinded to the results from the clinical examination will perform the ultrasound measurements. The physician responsible for the labor will be blinded to the ultrasound measurements.

Ultrasound examinations between contractions

Due to considerations described below, only one recording/acquisition will be performed of each of the following:

A) Head position B) Head-perineum distance C) Midline angle D) Angle of progression E) 3D sagittal transperineal acquisition In addition single scans are performed during active pushing as described under B) and D) (and a 3D sagittal scan when possible).

A) Head position Position will be assessed in 2D with a transabdominal scan as described by Akmal4 and 3D in a transperineal scan as described by Ghi et al22. Fetal head position will be recorded as a clock dividing the circle in 24 divisions

Positions ≥02.30 and ≤03.30 hours should be recorded as left occiput transverse and positions ≥08.30 and ≤09.30 as right occiput transverse. Positions >03.30 and <08.30 should be recorded as occiput posterior and positions >09.30 and <02.30 as occiput anterior.

Head-perineum distance will be assessed with transperineal ultrasound. The women will be examined lying flat (or almost flat) in bed with flexed hips and knees position. The bladder should be emptied immediately before the ultrasound examination.

Head-perineum distance will be measured as the shortest distance between the outer bony limit of the fetal skull and the perineum with a transabdominal transducer placed transperineally between the labia in a transverse view (posterior fourchette - posterior commissure of the labia minor)

Midline angle will be measured as described by Ghi22. In a transverse transperineal scan the angle between the midline of the fetal head and a sagittal line through the maternal pelvis will be measured. This recording will also be performed in a transverse scan.

Angle of progression will be measured as described by Barbera and Kalache as the angle between the long axis of the symphysis pubis and the tangent of the skull in a transperineal sagittal scan.

The following outcome variables will be recorded upon delivery Main outcome

* Time from start of vacuum assisted traction to delivery (the entire body is delivered) Secondary outcomes
* Number of contraction before delivery
* Number of cup detachments
* Successful/failed vaginal operative delivery
* Forceps applied/not applied
* Perineal tears
* APGAR score of newborn.
* Arterial umbilical cord blood pH and BD (base deficit) values.
* Position at delivery

Statistics:

The time interval between start of operative vaginal delivery and delivery will be evaluated for the fetal head-perineum distance and angle of progression using survival analyses (Kaplan-Meier analyses and Cox regression analyses).

Categorical variables will be analyzed using Chi-square test and Fischer exact test, and continuous variable will be analyzed using T-test or Mann-Whitney U-test.

The predictive values for a successful operative vaginal delivery will be evaluated using receiver-operating characteristics (ROC) curves. The area under the curve (AUC, - 95% CI) is considered to have discriminatory potential if the lower limit of the CI exceeded 0.5.

Ultrasound measurements, digital assessment of station and dilatation, induction of labor, maternal age, gestational age and birth weight will be analyzed in logistic regression analyses with vaginal delivery vs. cesarean section as dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* prolonged second stage of labour

Exclusion Criteria:

* Suspected asphyxia before the start of vacuum extraction

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Nulliparous women with a singleton live fetus in cephalic presentation at term (≥ 37 weeks) with prolonged active second stage and a clinical decision to expedite delivery by vacuum due to poor progression
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time from start of vacuum assisted traction to delivery | Active second stage of labor to1 hour after delivery
  The duration of a vacuum extraction will be measured. Therefore, the time frame is for this variable is only the second stage of labor. However, the time frame including all variables will be from the start of active second stage of labor - 1 hour after delivery.

SECONDARY OUTCOMES:
Successful/failed vaginal operative delivery (vaginal delivery vs. cesarean section | Active second stage of labour
  Successful or failed operative deliveries will be recorded. The time frame is also for this variable only the second stage of labor.

OTHER OUTCOMES:
Apgar score | first ten minutes after delivery
  Apgar score is assessed after 1,5 and 10 minutes
ph and base excess in umibical cord | first 5 minutes after delivery
  blood test from the umbilical board
birth weight and head circumference | First hour after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn M Eggebø, phd, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan WA, Eggebo TM, Ferguson M, Lees C. Simple two-dimensional ultrasound technique to assess intrapartum cervical dilatation: a pilot study. Ultrasound Obstet Gynecol. 2013 Apr;41(4):413-8. doi: 10.1002/uog.12316. PMID 23024020
- [Background] Tutschek B, Torkildsen EA, Eggebo TM. Comparison between ultrasound parameters and clinical examination to assess fetal head station in labor. Ultrasound Obstet Gynecol. 2013 Apr;41(4):425-9. doi: 10.1002/uog.12422. Epub 2013 Mar 14. PMID 23371409
- [Background] Torkildsen EA, Salvesen KA, VON Brandis P, Eggebo TM. Predictive value of ultrasound assessed fetal head position in primiparous women with prolonged first stage of labor. Acta Obstet Gynecol Scand. 2012 Nov;91(11):1300-5. doi: 10.1111/j.1600-0412.2012.01503.x. Epub 2012 Aug 22. PMID 22774859
- [Background] Torkildsen EA, Salvesen KA, Eggebo TM. Agreement between two- and three-dimensional transperineal ultrasound methods in assessing fetal head descent in the first stage of labor. Ultrasound Obstet Gynecol. 2012 Mar;39(3):310-5. doi: 10.1002/uog.9065. PMID 21630362
- [Background] Torkildsen EA, Salvesen KA, Eggebo TM. Prediction of delivery mode with transperineal ultrasound in women with prolonged first stage of labor. Ultrasound Obstet Gynecol. 2011 Jun;37(6):702-8. doi: 10.1002/uog.8951. Epub 2011 May 3. PMID 21308837
- [Background] Eggebo TM, Okland I, Heien C, Gjessing LK, Romundstad P, Salvesen KA. Can ultrasound measurements replace digitally assessed elements of the Bishop score? Acta Obstet Gynecol Scand. 2009;88(3):325-31. doi: 10.1080/00016340902730417. PMID 19172418
- [Background] Eggebo TM, Heien C, Okland I, Gjessing LK, Romundstad P, Salvesen KA. Ultrasound assessment of fetal head-perineum distance before induction of labor. Ultrasound Obstet Gynecol. 2008 Aug;32(2):199-204. doi: 10.1002/uog.5360. PMID 18528923
- [Background] Henrich W, Dudenhausen J, Fuchs I, Kamena A, Tutschek B. Intrapartum translabial ultrasound (ITU): sonographic landmarks and correlation with successful vacuum extraction. Ultrasound Obstet Gynecol. 2006 Nov;28(6):753-60. doi: 10.1002/uog.3848. PMID 17063455
- [Background] Kalache KD, Duckelmann AM, Michaelis SA, Lange J, Cichon G, Dudenhausen JW. Transperineal ultrasound imaging in prolonged second stage of labor with occipitoanterior presenting fetuses: how well does the 'angle of progression' predict the mode of delivery? Ultrasound Obstet Gynecol. 2009 Mar;33(3):326-30. doi: 10.1002/uog.6294. PMID 19224527
- [Background] Barbera AF, Pombar X, Perugino G, Lezotte DC, Hobbins JC. A new method to assess fetal head descent in labor with transperineal ultrasound. Ultrasound Obstet Gynecol. 2009 Mar;33(3):313-9. doi: 10.1002/uog.6329. PMID 19248000
- [Background] Eggebo TM. Ultrasound is the future diagnostic tool in active labor. Ultrasound Obstet Gynecol. 2013 Apr;41(4):361-3. doi: 10.1002/uog.12417. No abstract available. PMID 23641509
- [Background] Ghi T, Farina A, Pedrazzi A, Rizzo N, Pelusi G, Pilu G. Diagnosis of station and rotation of the fetal head in the second stage of labor with intrapartum translabial ultrasound. Ultrasound Obstet Gynecol. 2009 Mar;33(3):331-6. doi: 10.1002/uog.6313. PMID 19202576
- [Background] Ghi T, Youssef A, Maroni E, Arcangeli T, De Musso F, Bellussi F, Nanni M, Giorgetta F, Morselli-Labate AM, Iammarino MT, Paccapelo A, Cariello L, Rizzo N, Pilu G. Intrapartum transperineal ultrasound assessment of fetal head progression in active second stage of labor and mode of delivery. Ultrasound Obstet Gynecol. 2013 Apr;41(4):430-5. doi: 10.1002/uog.12379. PMID 23288706
- [Background] Youssef A, Maroni E, Ragusa A, De Musso F, Salsi G, Iammarino MT, Paccapelo A, Rizzo N, Pilu G, Ghi T. Fetal head-symphysis distance: a simple and reliable ultrasound index of fetal head station in labor. Ultrasound Obstet Gynecol. 2013 Apr;41(4):419-24. doi: 10.1002/uog.12335. Epub 2013 Mar 6. PMID 23124698